CLINICAL TRIAL: NCT05550727
Title: The PorchLight Project
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Lutheran Social Service of Minnesota (Unknown); Brown University (Other); The University of Texas at Arlington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00013917
Record Dates: First submitted 2022-08-08; First posted 2022-09-22 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Memory Loss; Alzheimer Disease; Dementia
MeSH Terms: conditions — Memory Disorders; Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PorchLight (Experimental)
  Interventions: Other: PorchLight
- Control (No Intervention)

INTERVENTIONS:
Other: PorchLight — The PorchLight Project intervention consists of three components: 1) CARES® Dementia Care Specialist online training modules; 2) a PorchLight Project training course; and 3) monthly check-in sessions.
  Arms: PorchLight

SUMMARY:
The proposed project is a fully embedded pragmatic trial (R01), following an R61 pilot collaboration with Lutheran Social Service of Minnesota (LSS-MN).

For this project: a) the training program for Senior Companions that was developed in the R61 Phase will now be delivered as part of a routine onboarding process provided by LSS-MN to all senior support volunteers in half of their program regions across Minnesota; LSS-MN will offer the PorchLight Project program to all regions and volunteers in the state during the final months of the proposed NIA project, consistent with quality improvement approaches; and b) LSS-MN will administer regular surveys to volunteers, clients, and caregivers as part of ongoing tracking and quality improvement efforts. The University of Minnesota investigators will not collect data nor administer training, as these activities will be fully integrated into the workflow of LSS-MN. [Note: Since it was learned that caregivers receiving services/affiliated with LSS-MN programming who receive surveys are for the most part not providing care to LSS-MN clients, as of fall 2024, UMN will no longer request and analyze data on LSS-MN caregivers.]

UNIVERSITY OF MINNESOTA INVOLVEMENT:

The University of Minnesota and collaborating investigators outside of LSS-MN will only 1) assist in survey item selection, 2) randomize the LSS-MN regions for the initial phases of the real-world trial for evaluation purposes, 3) analyze the de-identified data shared by LSS-MN, and 4) disseminate the project results in scientific, practice, and policy outlets/contexts.

ELIGIBILITY:
Inclusion Criteria:

In keeping with the incorporation of pragmatic design elements, the eligibility criteria of volunteers and persons with AD/ADRD is deliberately lax in order to best reflect LSS-MN "routine practice." Participants must be either a volunteer or client involved in the LSS-MN standard Caregiver & Companion Program service programs. Programmatic and survey data on the volunteers, clients, and proxies involved will be shared with the UMN team. While all data received may be analyzed (see analysis section below), data analysis is expected to focus on those who meet the following additional criteria:

* Volunteers who are listed in the LSS database.
* Clients with cognitive concerns (i.e. minor confusion, memory loss, diagnosis for their memory loss, or concerns about cognition) via the LSS-MN surveys and/or the LSS-MN CRM database.

If memory loss is indicated via the database or survey, it will be assumed that the client has memory loss, even if there are discrepancies. Due to the nature of the data, we expect discrepancies to exist and will document other decisions made during analysis.

Exclusion Criteria:

As data is made available, the UMN research team expects to receive survey data from all the clients and volunteers in LSS-MN Caregiver & Companion Services programming who complete the surveys, and those included in the LSS database. Since LSS-MN administers surveys to every client and volunteer involved in their LSS-MN Caregiver & Companion program (as able), data likely will be obtained from individuals who do not meet the memory-specific criteria. However, as needed, UMN may choose to exclude one or more of the following from analysis. Again, the researcher/research staff best judgement will be used when conducting analyses and will document decisions accordingly:

● Clients who do not have memory loss

In addition, any client and volunteer can choose to not complete surveys, so we would not have survey data from those individuals, and may continue with routine attempts at surveying at the next data collection time-point. Missing surveys may be considered during analysis.

Please note: Due to the eligibility criteria for volunteers and clients in the LSS-MN program, we do not anticipate any data for those under 18 years of age. Although the real-world, pragmatic design will allow us to include caregivers under the age of 21), it is important to note that LSS-MN's most recent data on caregivers participating in their volunteer programs indicate none under the age of 21

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in Volunteer Competence [Volunteers only] | Baseline, 6 months, and 12 months
  6-items assess the preparedness to provide visiting services for clients with a variety of conditions, including memory loss. This measure was designed for LSS-MN to determine the proportion of volunteers who indicate their level of preparedness.
Change in De Jong Gierveld Scale [Clients only] | Baseline, 6 months, and 12 months
  6-items assessing loneliness
Change in Patient-Reported Outcomes Measurement Information System Global Health Scale [All participants] | Baseline, 6 months, and 12 months
  10-items assessing physical health, mental health, and quality of life.

SECONDARY OUTCOMES:
Program Cost-Effectiveness | 12 months
  Incremental cost-effectiveness ratio (ICER) is the difference between the cost of the PorchLight Project and the usual LSS-MN Caregiver & Companion Services divided by the difference in the benefit (is the person with AD/ADRD's quality-adjusted life-years [QALYs]) between the PorchLight Project and the usual Caregiver & Companion Services.

OTHER OUTCOMES:
Change in Live Well at Home Rapid Screen [Clients only] | Baseline, 6 months, and 12 months
  6-items regarding falls, caregiving, living status, and cognition
Change in Experience/impact/satisfaction related to LSS programming [All participants] | Baseline, 6 months, and 12 months
  Experience/impact related to LSS programming (Volunteers: 3 quantitative, 3 open-ended items; Clients: 11 quantitative and 2 open-ended items. These items were designed for LSS-MN to assess both the proportion of participants who are satisfied with LSS programming, and to provide qualitative data about their experience.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota (with Lutheran Social Service of Minnesota), Minneapolis, Minnesota, United States